CLINICAL TRIAL: NCT02212496
Title: Identification the Cause of Cerebral Infarction in Patients With Cancer
Status: Completed | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Chin-Sang Chung, MD, PhD, Samsung Medical Center
Other Study IDs: 2014-07-136
Record Dates: First submitted 2014-08-06; First posted 2014-08-08 (Estimated); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Cryptogenic Embolic Stroke; Active Cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cancer-associated stroke: Cryptogenic embolic stroke with active cancer
- Cryptogenic embolic stroke: Cryptogenic embolic stroke without active cancer

SUMMARY:
Although there has been increasing interest in the association between cancer and cerebrovascular disease, the underlying pathophysiology of stroke in cancer patients is still not fully understood. The aim of this study is to investigate the stroke mechanisms in patients with cancer-associated stroke.

DETAILED DESCRIPTION:
Patients with cryptogenic embolic stroke will be prospectively enrolled and categorized into two groups according to the presence of active cancer: cryptogenic embolic stroke with active cancer (cancer-associated stroke) vs. without active cancer (cryptogenic embolic stroke). All patients will undergo brain MRI/MRA, 12-lead electrocardiography, transthoracic and transesophageal echocardiography with injection of agitated saline, and 24-hour Holter and/or telemonitoring. Duplex ultrasonography to detect venous thrombosis of the lower extremity will also be performed in patients with a positive right-to-left shunt on echocardiography.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with acute ischemic stroke who presented within 7 days from symptom onset
* Subjects who had embolic infarction outside the perforator territory revealed by diffusion-weighted imaging
* Subjects with undetermined cause of stroke despite of initial evaluation including electrocardiogram and brain imaging upon admission
* Subjects who performed brain magnetic resonance image (MRI) and MR angiography (MRA), cardiac work-ups (12-lead electrocardiography, transthoracic and/or transesophageal echocardiography with injection of agitated saline (or agitated saline transcranial Doppler monitoring), and 24-hour Holter and/or telemonitoring)
* Subjects with informed consent

Exclusion Criteria:

* Subjects with single subcortical infarction
* Subjects with primary brain tumor
* Inability to perform comprehensive studies
* Refusal or withdrawal of the consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Embolic stroke of undetermined source with or without cancer, admitted to Samsung Medical Center (tertiary hospital with comprehensive stroke and cancer center)
Sampling Method: Probability Sample
Enrollment: 118 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Prevalence of deep vein thrombosis and microembolic signal in cancer related stroke patients | Within one week after enrollment
  Venous thromboembolism was investigated via Doppler sonography and/or computed tomography pulmonary angiography combined with venous phase CT angiography of the lower extremities. Microembolic signal was detected via transcranial Doppler sonography on symptomatic cerebral circulation

SECONDARY OUTCOMES:
Impact of intravascular thrombosis on infarct volume | Within one week after enrollment
  Infarct volume was measured by diffusion-weighted MR imaging and apparent diffusion coefficient calculated from imaging data. Univariate and multivariate linear regression was performed in ESUS patients with cancer (adjusted for age, sex, overt DIC).
Impact of intravascular thrombosis on survival | Till the event of death occurs in enrolled patients
  Survival time (in years) was measured by subtracting admission date from the date the patient had expired. Cox proportional hazard analysis was used to evaluate association between intravascular thrombosis and survival (adjusted for age, sex, NIHSS, presence of overt DIC, infarct volume, metastasis, and histologic type).

CONTACTS AND LOCATIONS:
Overall Officials: Chin-Sang Chung, MD, PhD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Ha J, Lee MJ, Kim SJ, Park BY, Park H, Cho S, Chung JW, Seo WK, Kim GM, Bang OY, Chung CS. Prevalence and Impact of Venous and Arterial Thromboembolism in Patients With Embolic Stroke of Undetermined Source With or Without Active Cancer. J Am Heart Assoc. 2019 Nov 5;8(21):e013215. doi: 10.1161/JAHA.119.013215. Epub 2019 Oct 23. PMID 31640456